CLINICAL TRIAL: NCT06724432
Title: Evaluation of Effects of Melatonin in Reducing Postoperative Pain and Oxidative Stress in Children Undergoing Surgery,. Trought Circulating miR-34 and miR-124a, 4-Hydroxynonenal and Sirtuin 1 (SIRT1) Plasma Concentrations.
Brief Title: Analgesic and Antioxidant Effects of Melatonin in Pediatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Collaborators: University of Messina (Other); University of Florida (Other); University of Siena (Other); University of Urbino "Carlo Bo" (Other)
Responsible Party: Principal Investigator, Serafina Perrone, Professor, University of Parma
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ethics committee 125222022
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pain; Oxidative Stress Response
Keywords: children; surgery; postoperative pain; analgesia; melatonin; 4-hydroxynonenal (4-HNE); sirtuin 1 (SIRT1); miR-34; miR-124a
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: children were randomly assigned to oral supplementation with melatonin or placebo (5% dexstrose), before induction of an anesthesia for surgery
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin arm (Experimental): Mel treated children receive a single dose of oral melatonin 0.5 mg/kg (for a max 10 mg). Melatonin (Dicoson, Dicofarm, Italy) is prepared by a dedicated resident in a fixed volume of 5 mL by adding water to a syringe without a needle.
  Interventions: Drug: oral melatonin
- Control arm (Placebo Comparator): Children in the Control group receive 5 ml of 5% dextrose solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: oral melatonin — Melatonin treated children receive a single dose of oral melatonin 0.5 mg/kg (for a max 10 mg) in a fixed volume of 5 mL of water , 1 hour before induction of anesthesia for surgery
  Arms: Melatonin arm
Drug: Placebo — Children in the Control group receive 5 ml of 5% dextrose solution once 1 hour before induction of anesthesia
  Arms: Control arm

SUMMARY:
Background. Long-term consequences of postoperative pain are detrimental in children. We tested the hypothesis that melatonin reduces postoperative pain and oxidative stress involving sirtuin pathway in children undergoing surgery.

Methods. Thirty-one children were randomly assigned to oral supplementation with melatonin or placebo, before surgery. Plasma levels of 4-hydroxynonenal (4-HNE), melatonin, sirtuin 1 (SIRT1), and circulating miR-34 and miR-124a were analyzed at T0 (pre-hospitalization), T1 (before surgery), and T2 (1 h after the end of the surgery).

DETAILED DESCRIPTION:
Melatonin shows a potential role in protecting neonates undergoing surgery from the deleterious effects of oxidative stress (OS). After administration of exogenous melatonin, a significant reduction in lipid and protein peroxidation in the postoperative period has been reported in neonates. Recently, Song et al. reported that sirtuin 1 (SIRT1) also plays a critical role in the pathogenesis of pain, showing analgesic effects in chronic pain conditions such as neuropathic and inflammatory pain. In this prospective, randomized, double-blind pilot study, we test the hypothesis that melatonin reduces OS and postoperative pain involving the sirtuin pathway in children undergoing surgery.

Melatonin (Dicoson, Dicofarm, Italy, 5 drops = 1 mg) was administered orally. The product is listed in the Register of Dietary Supplements on the website of the Ministry of Health (http://www.ministerosalute.it/alimenti/dietetica) and is classified with the following code: 943314283. This product is subject to the European Directive on Foodstuffs according to DL n. 169 of May 21, 2004, and not to the European Directive on Medicines 2001/20/EC transposed at the Italian level with D.L. n. 211 of June 24, 2003. Melatonin administration has a good safety profile, with no known adverse effects.

Melatonin plasma levels were assessed at each experimental time point (T0, T1, T2) using a competitive enzyme-linked immunosorbent assay (cELISA) kit from Antibodies.com (A87093) according to the manufacturer's instructions. T1 and T2 plasma samples from Mel treated children suspected of containing concentrations higher than the highest standard (500 pg/mL) were diluted 1:100 (v/v) with sample diluent prior to analysis. Color development was monitored at 450 nm in a Thermo Scientific (MultiSkan FC) microplate reader, and a standard curve (range 7.813-500 pg/mL) was generated using a four-parameter logistic (4-PL) curve fit. The sensitivity of the assay was 4.688 pg/mL; the intra- and inter-assay coefficients of variation were <8% and <10%, respectively.

4-Hydroxynonenal (4-HNE) as a marker of lipid peroxidation was measured to evaluate OS by using a cELISA kit from Antibodies.com (A86962). Plasma concentrations were calculated by reading the absorbance at 450 nm and referring to the standard curve (range 31.25-2000 pg/mL). The sensitivity of the assay was 18.75 pg/mL; the intra- and inter-assay coefficients of variation were <8% and <10%, respectively.

SIRT1 was quantified using an ELISA kit from Invitrogen (EH427RB). Plasma samples were diluted 1:2 as indicated by the Manufacturer before analysis. SIRT1 concentrations were calculated by absorbance reading at 450 nm and referring to the standard curve (range 1.23-300 ng/mL). The sensitivity of the assay was 1.23 ng/mL; the intra- and inter-assay coefficients of variation were <10% and <12%, respectively.

We performed microRNA analyses based on the quali-quantitative plasma sample available (N=3 at each time point, T0, T1, and T2). MicroRNAs (miR-34 and miR-124a) were isolated from plasma using the Norgen total RNA isolation kit13.The Plasma microRNAs and spike-in cel-miR-39 expressions were evaluated using the TaqMan miRNA assay. The TaqMan miRNA reverse transcription kit was used to reverse transcribe miRNAs. Subsequently, RT-qPCR was performed in 20 μL of PCR mix containing 1 μL of 20× TaqMan miRNA assay, which contained PCR primers and probes (5'-FAM), 10 μL of 2×TaqMan Universal PCR Master Mix No Amp Erase UNG and 5 μL of reverse-transcribed product. The reaction was first incubated at 95 °C for 10 min followed by 40 cycles at 95 °C for 15 s and at 60 °C for 1 min. The quantitative real-time PCR (RT-qPCR) was performed on a ABIPRISM 7500 Real Time PCR System. Data was analyzed by a 7500-system software (1 1.4.0) with the automatic comparative threshold (Ct) setting for adapting baseline. Detection thresholds were set at 35 Ct. The relative amounts of miR-34 and miR-124a were calculated using the Ct method: ΔCt = Ct (miR-34/miR-124a) - Ct (refence miRNA); 2-ΔCt.

ELIGIBILITY:
Inclusion Criteria:

Children between 3 and 5 years of age scheduled for elective surgery, parental consent

Exclusion Criteria:

Children with cerebral malformations and/or injuries, or surgery in the afternoon or at night to eliminate conditions that could affect melatonin production, or denial of parental consent

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Plasma levels evaluation of 4-hydroxynonenal (4-HNE), melatonin, sirtuin 1 (SIRT1), and circulating miR-34 and miR-124a | Samples of 0.2 mL of plasma were collected at T0 (pre-hospitalization, 1 day before surgery), T1 (before surgery, pre-anesthesia) and T2 (at 1 h after the end of the surgery and awakening after anesthesia), and biochemical analyses performed.
  Melatonin plasma levels were assessed using a competitive enzyme-linked immunosorbent assay (cELISA) kit from Antibodies.com (A87093) according to the manufacturer's instructions.
  4-Hydroxynonenal (4-HNE) as a marker of lipid peroxidation was measured to evaluate OS by using a cELISA kit from Antibodies.com (A86962).
  SIRT1 was quantified using an ELISA kit from Invitrogen (EH427RB). MicroRNAs (miR-34 and miR-124a) were isolated from plasma using the Norgen total RNA isolation kit13.The Plasma microRNAs and spike-in cel-miR-39 expressions were evaluated using the TaqMan miRNA assay.

SECONDARY OUTCOMES:
control post operative pain in children treated with melatonin compared to placebo | 48 hours after surgery were considered as post-operative period
  doses of paracetamol to control post operative pain were recorded in children treated with melatonin compared to placebo

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University Hospital of Messina, Italy, Messina
  - Neonatology Unit, Department of Medicine and Surgery, University of Parma, Pietro Barilla Children's Hospital, Parma

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT06724432/Prot_SAP_000.pdf